CLINICAL TRIAL: NCT05271266
Title: A Multicenter, Prospective, Non-interventional Cohort Study to Evaluate the Safety and Treatment Pattern of Sodium Zirconium Cyclosilicate for Hyperkalaemia Management in Real World Practice in China
Acronym: ACTUALIZE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9483R00001
Record Dates: First submitted 2022-01-13; First posted 2022-03-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hyperkalaemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — This study is a non-interventional study and will not collect the biospecimen.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a multi-center prospective (primary data) non-interventional cohort study which enrolls 1500 patients including new and ongoing users on SZC at Study Enrollment Day in real-world clinical practice. The eligible study patients will be identified by physicians in each study site by assessing the patients or reviewing the medical record.

The prescription (including initiation, dose-adjusting or interruption) or discontinuation of SZC will be determined by physicians as per real-world clinical practice and in accordance with the local label. Any AZ employee, or member of the research operation team must not intervene in the decision-making of any physician or patient through any approach, at any time during the study.

Every patient will be followed up according to standard clinical practice for 6 months from enrolment.

DETAILED DESCRIPTION:
Background/Rationale:

Hyperkalaemia (HK) is a common electrolyte disturbance in clinical practice, defined as serum potassium (sK) beyond the normal range. The cut-off value for HK diagnosis is 5.0 mmol/L in most international guidelines[1, 2]. HK changes potassium ion gradient across the cell membrane and affects the excitability and conductivity of cardiomyocytes, leading to various types of arrhythmias, including ventricular arrhythmia, cardiac arrest and sudden death[3]. In the general population, the prevalence of HK is about 2-3%[4-6]. In an epidemiological survey among outpatients in China, 3.86% of general outpatients experienced HK, and the proportion of patients who experienced HK increased in patients with chronic kidney disease (CKD), heart failure, diabetes and hypertension [7].

Sodium Zirconium Cyclosilicate (SZC) is a non-absorbed, non-polymer inorganic powder with a uniform micropore structure that preferentially captures potassium in exchange for hydrogen and sodium cations. SZC captures potassium throughout the entire gastrointestinal (GI) tract and reduces the concentration of free potassium in the GI lumen, thereby lowering sK levels and increasing faecal potassium excretion to resolve HK[8].

The potassium-lowering effects of SZC have been demonstrated in three randomised, double-blind, placebo-controlled trials in patients with HK [9-11]. In addition, two open-label maintenance studies tested long-term safety of SZC[12, 13]. These five studies included 1,760 patients given doses of SZC; 507 exposed for at least 360 days. In the studies, SZC reduced sK and maintained normal sK levels regardless of the underlying cause of HK, age, sex, race, comorbid disease or concomitant use of renin-angiotensin and aldosterone system inhibitors (RAASi).

As of 21 September 2019, the data cut-off date, approximately 2,580 patients have been cumulatively exposed to SZC in completed and on-going clinical trials. Based on the data available now, oedema-related events (including fluid overload, fluid retention, generalised oedema, hypervolaemia, localised oedema, oedema, oedema peripheral, peripheral swelling) and hypokalemia are common (frequency ≥1/100 to >1/10) adverse reactions reported with SZC.

In December 2019, SZC was approved in China. It is indicated for the treatment of HK in adults. According to the National Medical Products Administration (NMPA) Regulations, the safety profile of a newly approved drug should be intensively monitored within 5 years from the date of first approval for import. As compared with the pre-market phase II/III studies, post-market real world observational studies can observe the product safety profile in a broader population and reflect the situation in routine clinical practice, which can meet the request of the Guidelines of Drug Intensive Monitoring of Manufacturers. This study is expected to enhance and supplement currently available SZC safety and tolerability data with expansion to broader Chinese population.

Objectives:

Primary objectives: To describe the safety and tolerability of SZC for hyperkalemia management in Chinese patients in terms of adverse events (AEs), serious adverse events (SAEs) and discontinuations of SZC due to adverse events (DAEs), and specific AEs (oedema and hypokalemia).

Secondary objectives:

* To describe the safety and tolerability of SZC for HK management in Chinese hyperkalaemic patients in terms of AEs, SAEs and DAEs, and specific AEs (oedema and hypokalemia) judged by the study investigators to be causally related to SZC.
* To understand the treatment pattern of SZC in real-world clinical practice for treating HK in Chinese patients.
* To describe the sK level of patients treated with SZC during the observational period

Methods:

Study design: The study is a multi-center prospective observational cohort study which will enroll patients who are ongoing and new users for HK management on SZC at study enrolment in real-world clinical practice. The eligible patients will be identified by physicians in each study site by assessing the patients or reviewing the medical record.

The prescription (including initiation, dose-adjusting or interruption) or discontinuation of SZC will be determined by physicians as per real-world clinical practice and in accordance with the local label. Any AZ employee, or member of the research operation team will not intervene the decision-making of any physician or patient through any approach, at any time during the study.

Every patient will be followed up according to standard clinical practice for 6 months from enrolment.

At Study Enrollment Day (Day 1) the patients will be classified into 2 groups as new user group and ongoing user group. New users are defined that the patients without SZC treatment within 7 days before enrollment take SZC on Study Enrollment Day. Ongoing users are defined that the patients with SZC treatment within 7 days before Study Enrollment Day continue SZC treatment after enrollment. The patients with previous SZC treatment who will not continue taking SZC treatment after enrollment will not be included.

Per standard clinical practice, new users of SZC should visit doctors within 1-3 days after initiation of treatment for potassium re-testing, while ongoing users should visit doctors once every 1-2 month for potassium monitoring or chronic disease consultation.

For new user group

* The "study index SZC treatment episode" starts at Study Enrollment Day.
* Follow-up visits will be planned on the 3rd day, the 1st month, the 3rd month and the 6th month from Study Enrollment Day.

For ongoing user group

* The "study index SZC treatment episode" started prior Study Enrollment Day.
* Follow-up visits will be planned on the 1st month, the 3rd month and the 6th month from Study Enrollment Day.

Visits of Day 1 (Study Enrolment Day) and Day 3 (only applicable for patients in new user group) are onsite. For visits at Month 1, Month 3 and Month 6, if the patient continues taking SZC treatment at the visit time points, his/her visit will be onsite. Otherwise, the visit will be conducted by phone-call. At each visit, safety outcomes, sK measurements data (if available), treatment data of SZC (as applicable) and other related data (if available) will be collected, as detailed in Section 6.1.2.

Data Source: This study will be based on primary (prospective) data collected from approximately 60 hospitals in China recruiting 1500 patients. The site investigators will be responsible for ensuring that all the required data are collected and entered into the electronic case report form (eCRF).

Study Population: This study will enroll Chinese patients who are new and ongoing users of SZC defined above at Study Enrolment Day. Eligible patients can be those under or not dialysis treatment.

Exposure: Drug exposure of SZC treatment. Treatment dose and duration of SZC is at the discretion of the patient's treating physician.

Outcome (s): Study measures will be collected at Study Enrollment Day (Day 1) and at the scheduled study visits.

Primary Endpoints:

Occurrence of AEs, SAEs and DAEs, specifically AEs (oedema and hypokalemia). Oedema is defined as an AE with one of the following preferred terms (PTs): Includes Fluid overload, Fluid retention, Generalised oedema, Hypervolaemia, Localised oedema, Oedema, Oedema peripheral, Peripheral swelling. Hypokalemia is defined as an AE with laboratory potassium value test below 3.5 mmol/L

Secondary Endpoints:

* Occurrence of AEs, SAEs and DAEs, specifically AEs (oedema and hypokalemia), judged by the investigators to be causally related to SZC.
* Average SZC daily dosage, frequency of different SZC dosages, duration of SZC treatment, dose changes and reasons for any dose changes.
* Change in sK tested between V1 and V3, as well as average (within patient) sK levels during the study. An evaluation of whether or not a patient tends to be normokalemic. Two criteria for normokalemia will be considered:

  * sK between 3.5 to 5.0 mmol/L, inclusive
  * sK between 3.5 to 5.5 mmol/L, inclusive. Sample Size Justification: The total sample size for this study is 1500 according to the mandatory request by NMPA. It's assumed that the size of new users group will be ranging from 500 to 1000, while the rest would be ongoing users group. Primary outcome measures will be: 1) Percentage of overall AEs, SAEs, DAEs and specific AEs (oedema and hypokalemia) during the first period (the time span between the first and the second visits after SZC is initiated, only include new users group); and 2) Incidence rates of overall AEs, SAEs, DAEs and specific AEs (oedema and hypokalemia) during second period (starting after the initial treatment period is over, include ongoing users group and possibly a subset of new users group). Detailed definition of first and second period will be provided in statistical analysis section.

For percentage of overall AEs, assuming the point estimate would be 10%, the assumed size of 500 to 1000 new users could provide the 95% confidence interval (CI) estimation from [7.4%, 12.6%] to [8.1%, 11.9%].

For incidence rates of overall AEs, assuming the point estimate would be 107.88 per 100 person-years, the assumed size of 500 to 1000 patients over 0.5 to 1.5 months could provide the 95% confidence interval from [71.32, 163.12] to [91.13, 127.72].

Sample size estimation under other scenarios as well as detailed description of estimation approach will be provided in section 5.4.

Statistical Analysis:

This study is primarily of descriptive character with no formal hypothesis testing for the objectives. The analyses will, as a rule, consist of estimates (of probabilities, rates, means, etc.), with the corresponding 95% CIs, as well as supportive descriptive statistics such as mean, standard deviation (SD), median, minimum, maximum, and quartiles.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year-old
* Provision of patient informed consent prior to any study procedure
* HK (sK+ > 5.0 mmol/L) diagnosed by physicians within 1 year before Study Enrolment Day
* Currently taking SZC, or has been prescribed and agree to start taking SZC since Study Enrolment Day.

Exclusion Criteria:

* Being unable to comply with study-specified procedures
* Has ever participated in current study before, or participating in any interventional study at Study Enrolment Day or within the last 3 months before Study Enrolment Day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll eligible Chinese patients who are new and ongoing users on SZC at Study Enrollment from approximately 60 sites in China recruiting 1500 patients. New users are defined that the patients without SZC treatment within 7 days before Study Enrollment Day take SZC treatment on Study Enrollment Day. Ongoing users are defined that the patients with SZC treatment within 7 days before Study Enrollment Day continue SZC treatment after enrollment. The patients with previous SZC treatment who will not continue taking SZC treatment after enrollment will not be included.
  Eligible patients will be those who meet all inclusion criteria but not any exclusion criteria. Eligible patients can be patients with or without hemodialysis treatment.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Safety laboratory tests associated with AEs, SAEs and DAEs, specifically AEs | From enrollment to the 6th month after Enrollment
  Serum electrolytes values（mmol/L）, serum BUN（mmol/L）, serum bicarbonate（mmol/L）, and others
The percentage of signs and symptoms associated with AEs, SAEs and DAEs, specifically AEs | From enrollment to the 6th month after Enrollment
  The percentage of edema, constipation and others

SECONDARY OUTCOMES:
Safety laboratory tests associated with AEs, SAEs and DAEs, specifically AEs | From enrollment to the 6th month after Enrollment
  Serum electrolytes values（mmol/L）, serum BUN（mmol/L）, serum bicarbonate（mmol/L）, and others
The percentage of signs and symptoms associated with AEs, SAEs and DAEs, specifically AEs | From enrollment to the 6th month after enrollment
  The percentage of edema, constipation and others
Medication information | From enrollment to the 6th month after enrollment
  SZC dosage(g), etc

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Lin, Doctor, Study Chair — The First Affiliated Hospital of Dalian Medical University
Locations (27):
- China (27):
  - Research Site, Anshan
  - Research Site, Beijing
  - Research Site, Benxi
  - Research Site, Changsha
  - Research Site, Changshu
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Handan
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jiaxing
  - Research Site, Kunshan
  - Research Site, Linfen
  - Research Site, Nanjing
  - Research Site, Nanyang
  - Research Site, Ningbo
  - Research Site, Qidong
  - Research Site, Shijiazhuang
  - Research Site, Shiyan
  - Research Site, Taian
  - Research Site, Taishing
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Xi'an
  - Research Site, Xinghua

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Shen N, Meng Q, Zhang L, Xie H, Zhao J, Xing C, Zuo L, Long G, Zhu Q, Shan C, Cai X, Yang J, Luo X, Wang J, Ye J, Wan X, Tian S, Wu Y, Lin Y, Yu X, Li Q, Liu X, Shi Z, Zhou J, Liu C, Cao Y, Wang N, Jiang X, Wu H, Hu Y, Li L, Wang Z, He J, Cao J, Wu F, Ma C, Yin X, Li Z, Wang H, Lin H. Evaluation of safety, effectiveness and treatment patterns of sodium zirconium cyclosilicate in management of hyperkalaemia in China: a real-world study protocol. BMJ Open. 2023 Mar 8;13(3):e070530. doi: 10.1136/bmjopen-2022-070530. PMID 36889826
- See also: D9483R00001_Redacted_CSR_Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9483R00001&attachmentIdentifier=dd80c741-8353-4e07-a716-a31fc7e76951&fileName=D9483R00001_Redacted_CSR_Synopsis.pdf&versionIdentifier=